CLINICAL TRIAL: NCT05307250
Title: M-Suubi: A Multi-Level Integrated Intervention to Reduce the Impact of HIV Stigma on HIV Treatment Outcomes Among Adolescents Living With HIV in Uganda
Brief Title: M-Suubi: A Multi-Level Integrated Intervention to Reduce the Impact of HIV Stigma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Fred Ssewamala, Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R01MH126892 (NIH)
Record Dates: First submitted 2021-12-21; First posted 2022-04-01 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: HIV/AIDS
Keywords: AIDS PREVENTION; ADOLESCENT; ADHERENCE; AIDS/HIV PROBLEM
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment Arm 1 (Experimental): Multiple Family Groups for HIV stigma reduction (MFG-HIVSR) plus FEE
  Interventions: Behavioral: Multiple Family Groups for HIV stigma reduction (MFG-HIVSR) plus FEE; Other: Bolstered Standard of Care (BSOC)
- Treatment Arm 2 (Experimental): Multiple Family Groups for HIV stigma reduction (MFG-HIVSR) plus FEE plus Group-based stigma reduction for educators (GED-HIVSR)
  Interventions: Behavioral: Multiple Family Groups for HIV stigma reduction (MFG-HIVSR) plus FEE plus Group-based stigma reduction for educators (GED-HIVSR).; Other: Bolstered Standard of Care (BSOC)
- Control Arm (Other): Bolstered Standard of Care (BSOC)
  Interventions: Other: Bolstered Standard of Care (BSOC)

INTERVENTIONS:
Behavioral: Multiple Family Groups for HIV stigma reduction (MFG-HIVSR) plus FEE — In addition to the BSOC, ALHIV and their caregivers will participate in a family strengthening intervention plus a family economic empowerment intervention.
  MFG is an evidence-based family-centered, group-delivered, evidence-informed, strength-based 10-session (weekly) intervention for children whose families struggle with poverty. Six additional sessions covering HIV stigma stigma-related issues will be added.
  ALHIV will receive a YDA with a 1:1 matched savings program at a financial institution accredited by the Bank of Uganda. Each YDA will be opened in the name of the adolescent, with their primary caregiver as a co-signer, until the adolescent turns 18 years. The account will then be matched with money from the program on 1:1 rate.
  Arms: Treatment Arm 1
Behavioral: Multiple Family Groups for HIV stigma reduction (MFG-HIVSR) plus FEE plus Group-based stigma reduction for educators (GED-HIVSR). — In addition to BSOC and MFG-HIVSR+FEE, ALHIV in this arm will receive the school-level HIV stigma reduction intervention targeting teachers, school nurses, matrons, and administrators (headteachers, director of studies) in their schools. GED-HIVSR seeks to impart educators in the intervention schools with HIV related knowledge, provide a safe space for educators to explore their personal values and bias that may promote or hinder their role of supportive individuals and systems for ALHIV, and empower them with knowledge and skills to act as change agents within their schools.
  Arms: Treatment Arm 2
Other: Bolstered Standard of Care (BSOC) — All participants (in control and treatment arms) will receive medical and psychosocial support as part of the BSOC. 1) Medical SOC: All public clinics, including our study sites, follow procedures for pediatric ART initiation and monitoring, as outlined in the National Department of Health Guidelines for pediatric HIV care in Uganda. Specifically, immediately after initiation, or if clinically unstable, ALHIV are seen more frequently (weekly to monthly). Laboratory data (VL and CD4 counts) are collected every six months until the patient is stabilized and then annually, using the National Health Laboratory Service standardized protocol. A

SUMMARY:
M-Suubi, a three arm cluster randomized study will examine the effects and cost-effectiveness of a multi-level intervention on HIV viral suppression among 840 adolescents living with HIV (ALHIV) enrolled in 42 secondary schools with a boarding section. The investigators will test the effects of a group-based HIV stigma reduction intervention for educators (GED-HIVSR), over and above the effects of multiple family groups with HIV stigma reduction combined with family economic empowerment (MFG-HIVSR plus FEE), relative to Bolstered Standard of Care (BSOC). ALHIV will be randomized at the school level to one of three study arms

DETAILED DESCRIPTION:
HIV stigma remains a formidable barrier to HIV treatment adherence among adolescents in Uganda, contributing to low rates of medication adherence and viral suppression (less than 50%) and high attrition from HIV treatment services. ALHIV experience HIV stigma (internalized, anticipated and enacted) in various settings, including families and schools, the most important developmental contexts that should otherwise be supportive of their development and wellbeing. One of the unique features about education in Uganda and other countries in Sub-Saharan Africa is the high proportion (over 60%) of school-going adolescents enrolled in boarding secondary schools - which represent a form of parental opt-in institutionalized care. ALHIV in schools are more disadvantaged and have lower levels of HIV treatment adherence due to high levels of HIV stigma within schools, rigid school structures and routines, lack of adherence support and food insecurity. Within families, HIV stigma is perpetuated in various forms including discrimination and violence, often due to unfounded fears of infection-hence undermining the quality of family relations and supports for ALHIV. Building on our research and current evidence on HIV stigma reduction, the investigators propose a multi-level three-arm cluster randomized study (M-Suubi) with the following specific aims: Aim 1: Examine the impact of M-Suubi on HIV viral suppression (primary outcome); and adherence to HIV treatment (keeping appointments, pharmacy refills, pill counts), and retention in care (secondary outcome); Aim 2: Examine the effect of M-Suubi on HIV stigma (internalized, anticipated and enacted), with secondary analyses to explore hypothesized mechanisms of change (e.g. depression) and intervention mediation; Aim 3: Assess the cost and cost-effectiveness of each intervention condition; and Aim 4: Qualitatively examine: a) participants' experiences with HIV stigma, HIV treatment adherence, and the intervention; and 2) educators' attitudes towards ALHIV, experiences with GED-HIVSR, and program/policy implementation post-training. The study will enroll 840 ALHIV recruited from 42 schools located within the greater Masaka region, heavily affected by HIV (prevalence 12% vs 7.3% national average). M-Suubi will be provided for 20 months, with assessments at baseline, 12, 24 and 36 months. Findings may inform combination intervention efforts to optimize HIV treatment outcomes and engagements in care among ALHIV.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive adolescents confirmed by medical report
* Prescribed antiretroviral therapy
* Enrolled in primary and secondary schools in a boarding section
* Caregivers of ALHIV who agree to participate in the study
* Teachers, school nurses, and administrators in the target schools who agree to participate in the study

Exclusion Criteria:

- A significant cognitive impairment that interferes with the participant's understanding of the informed consent process, or inability/unwillingness to commit to completing the study

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1851 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change HIV viral suppression | Baseline 12, 24 and 36 month follow-up
  Change in viral suppression will be assessed using viral load (VL) data collected from health clinic records. VL will be dichotomized between undetectable /suppression (VL< 40 copies/ml) and detectable/failed viral suppression (VL > =40 copies/ml) levels at each assessment time.

SECONDARY OUTCOMES:
Change in Adherence and retention in care | Baseline 12, 24 and 36 month follow-up
  Change in adolescent Self reported medication adherence. This will be measured using the Adherence and retention in care questionnaire focusing on the pharmacy refills, pill counts and missed appointments at each assessment time.
HIV Stigma Measure for Children | Baseline 12, 24 and 36 month follow-up
  HIV-associated stigma for children will be measured using the HIV Stigma Measure. We will measure the mean score over time. The total score range between 40- 160 with a high score indicating higher levels of perceived HIV-associated stigma.
The Shame Questionnaire for Children | Baseline 12, 24 and 36 month follow-up
  Shame related to living with HIV will be measured using the Shame Questionnaire. We will measure the mean score over time. The total score range between 0 and 16 with a higher score indicating higher levels of HIV-associated shame.

OTHER OUTCOMES:
Child Depression Inventory (CDI) | Baseline 12, 24 and 36 month follow-up
  Depressive Symptoms will be measured using the Child Depression Inventory (CDI) scale. We will measure the mean score on the CDI scale over time. The total score range between 0 and 28 with a high score indicating higher levels of depressive symptoms.
Post-Traumatic Stress Disorder (PTSD) | Baseline 12, 24 and 36 month follow-up
  Post-Traumatic Stress Disorder (PTSD) will be measured using the Child PTSD Reaction Scale. We will measure the mean score on the Child PTSD Reaction Scale over time. The total score range between 0 and 120, with a high score indicating higher levels of PTSD.
Tennessee Self-Concept Scale (TSCS) | Baseline 12, 24 and 36 month follow-up
  Self concept will be measured using the Tennessee Self-Concept Scale (TSCS). We will measure the mean score on the TSCS over time. The total score range between 20 and 100 with a high score indicating higher levels of self-concept.
Beck Hopelessness Scale (BHS) | Baseline 12, 24 and 36 month follow-up
  Hopelessness will be measured using the Beck Hopelessness Scale (BHS). We will measure the mean score on the BHS over time. The total score range between 0 and 20 with a high score indicating higher levels of hopelessness.
HIV Adherence Self-Efficacy Scale | Baseline 12, 24 and 36 month follow-up
  Self reported medication adherence will be measured by the number of times a child missed taking medication in the past 30 days, and number of days took medication the way they were supposed to.
  HIV Adherence Self-Efficacy Scale (HIV-ASES)
Family relations | Baseline 12, 24 and 36 month follow-up
  Change in family relations will be measured by Family Environment Scale
Social Support Behaviors Scale | Baseline 12, 24 and 36 month follow-up
  Social support from family members and friends will be measured using the Social Support Behaviors Scale (SSBS). We will measure the mean score on the SSBS over time. The total score ranges between 45-225, with higher score indicating higher levels of social support.
Rosenberg Self-Esteem Scale | Baseline 12, 24 and 36 month follow-up
  Self- Esteem will be measured using the Rosenberg Self-Esteem Scale. The total score range 0-30 where a score less than 15 may indicate a problematic low self esteem.
Savings Deposits | Baseline 12, 24 and 36 month follow-up
  Change in savings will be measured by Bank statements and financial diaries. Minimum savings will be 0.
Financial Literacy | Baseline 12, 24 and 36 month follow-up
  Change in Financial Literacy knowledge
Caregiver mental health | Baseline 12, 24 and 36 month follow-up
  Hopkins Symptom Checklists will be used to measure symptoms of anxiety and depression. We will measure the mean score of the Hopkins Symptoms Checklists over time. High score indicates severe levels of anxiety and depression.

CONTACTS AND LOCATIONS:
Locations (1):
- International Center for Child Health and Development Field Office, Masaka, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Once all of the data has been de-identified, cleaned, and validated, and main findings have been published, the Investigators expect to share data with the scientific community. The research team will make datasets available to any individual who makes a direct request to the PI and indicates the data will be used for the purposes of research (per Code of Federal Regulations Title 45 Part 46: "Research is defined as a systematic investigation, including research development, testing and evaluation, designed to develop or contribute to generalizable knowledge."). In sharing participant data, the team will follow Washington University in St. Louis' Office of Sponsored Projects' data sharing agreement.
Supporting Information: Study Protocol, Analytic Code

REFERENCES:
- [Derived] Mutumba M, Ssewamala FM, Nabunya P, Nattabi J, Namirembe R, Matovu F, Namatovu P, Mwebembezi A. HIV-related stigma and academic outcomes: the mediating role of mental health among adolescents living with HIV in Uganda. AIDS Care. 2025 Dec 29:1-12. doi: 10.1080/09540121.2025.2606202. Online ahead of print. PMID 41457981
- [Derived] Mutumba M, Ssewamala F, Namirembe R, Sensoy Bahar O, Nabunya P, Neilands T, Tozan Y, Namuwonge F, Nattabi J, Acayo Laker P, Mukasa B, Mwebembezi A. A Multilevel Integrated Intervention to Reduce the Impact of HIV Stigma on HIV Treatment Outcomes Among Adolescents Living With HIV in Uganda: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Oct 5;11(10):e40101. doi: 10.2196/40101. PMID 36197706